CLINICAL TRIAL: NCT00454948
Title: Home Based Nutrition Intervention Nad Play Group Exercise for Low-income Latinas
Brief Title: Nutrition Intervention and Play Group Exercise for Low-income Latinas
Acronym: CHICOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01DK073377-01 (NIH)
Record Dates: First submitted 2007-03-29; First posted 2007-04-02 (Estimated); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Obesity
Keywords: Obesity prevention; Dietary intake; Physical activity; Mexican American; Family Characteristics
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Home based Nutrition and Physical Activity (Experimental): Home-based nutrition sessions and park play activity sessions
  Interventions: Behavioral: Home-based nutrition sessions and play group exercise
- Group Nutrtion (Active Comparator): Group based nutrition classes and activity booklets
  Interventions: Behavioral: Group-based nutrition sessions and mail-out activities

INTERVENTIONS:
Behavioral: Home-based nutrition sessions and play group exercise
  Arms: Home based Nutrition and Physical Activity
Behavioral: Group-based nutrition sessions and mail-out activities
  Arms: Group Nutrtion

SUMMARY:
Obesity among Mexican-American women has the potential to become a public health crisis. Hispanics are one of the fastest growing minority populations in the United States and the prevalence of obesity in Mexican American woman is increasing at an alarming rate. Poor dietary practices, especially food habits that are acquired as families acculturate to the American food supply, and lack of exercise are thought to be associated with women's excess weight gain. Accordingly, interventions are needed to improve the dietary intake and physical activity levels of Mexican-American families.

We propose to conduct a randomized clinical trial in which women are randomly assigned to receive either family-based behavioral counseling (FBC) sessions and play group physical activity sessions or group based nutrition and exercise classes and health related activity worksheets to complete with their child. The FBC sessions, conducted by community health advisors, will use photographs of the family's food practices, taken by mothers, as visual aids in the counseling sessions. The control intervention will consist of group sessions using curricula designed to motivate women to exercise and to promote the Food Guide Pyramid recommendations using traditional Mexican-American foods. The primary outcome of the trial is mother's BMI. The secondary outcomes are dietary intake, moderate to vigorous physical activity and household food supplies. We hypothesize that within a one year time frame, women who are exposed to the FBC will have lower BMI's compared to women who receive the active placebo control intervention. The mechanisms through which we intend to change weight status are altering the type of foods purchased and cooking practices and promoting mothers to engage in physical activities with their children during their play. Measurements of secondary outcomes include three 24 hour dietary recalls, a household food inventory and activity monitoring using MTI actigraph monitors. In addition, mothers' reports of household food security level, and food purchase motives, will be collected as covariates. Measurements will be collected within one month of completing the interventions and at six months and one year follow-up.

DETAILED DESCRIPTION:
We propose to evaluate a family-based intervention designed to prevent obesity by increasing fruit and vegetable (F&V) intake, decreasing fat intake and increasing physical activity. The target group for the intervention is low-income Mexican-American mothers of preschool aged children. The intervention uses family-based behavioral counseling (FBC) sessions with a community health advisor (CHA) to promote changing the types of foods that mothers prepare and consume, and increasing the time that mothers spend being active with their children. In previous research, we have used this approach to improve Mexican-American school aged children's nutritional status. The mothers of these children were extremely motivated to improve their children's diets, and in doing so, improved their own health behaviors and reduced their BMI's. Accordingly, in the proposed research, we will conduct a randomized controlled trial with a sample of 250 Mexican-American mothers-child dyads to evaluate a family based intervention designed to prevent obesity in low income Mexican-American women. As families enroll in the study, they will be randomly assigned to either the FBC sessions or an active placebo control condition. Data will be collected immediately prior to participation in the intervention, within one-month of completing the intervention and at six months and one year follow-up. Mother's body mass index (BMI) will serve as the primary outcome variable. Multiple 24-hour dietary recalls, a modified household food inventory and physical activity monitoring will be used as secondary indices of program efficacy. The following hypotheses will be examined in this experiment.

Primary Hypothesis Women who receive the FBC sessions will have significantly lower BMI one year after randomization into the intervention compared to women whose families receive an active placebo control.

Secondary Hypotheses

Women who receive the FBC sessions will have significantly lower fat intakes and higher fruit and vegetable intakes, as measured by 24 hour recalls, one year after randomization into the intervention compared to women whose families receive an active placebo control.

Women who receive the FBC sessions will have significantly fewer high fat foods and significantly more fruits and vegetables in their homes, as measured by targeted household food inventories, one year after randomization into the intervention compared to women whose families receive an active placebo control.

Women who receive the FBC sessions will be significantly more active one year after randomization into the intervention, as measured by activity monitoring, compared to women whose families receive an active placebo control.

ELIGIBILITY:
Inclusion Criteria:

* Mother is of Mexican descent
* Mother has a child between the ages of 3 and 4.9 years

Exclusion Criteria:

* Child is eligible for kindergarten in the upcoming 6 months
* Mother is pregnant
* Mother is less then 4 months post partum
* Family plans on moving outside of San Jose in the upcoming 6 months
* Family shares food supplies with more than one other household
* Mother has medical condition or takes medication that affects weight
* Child has medical condition or takes medication that affects weight or growth

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2007-03; Primary Completion 2008-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
BMI at one year after randomization

SECONDARY OUTCOMES:
BMI percentile score of children one year after intervention
Dietary intake of mothers and their child one year after intervention as measured by multiple 24 hour recalls
Physical activity of mother and their child as measured by actigraph monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Donna M Matheson, PhD, Principal Investigator — Stanford University
Locations (1):
- San Jose, California, United States